# STATISTICAL ANALYSIS PLAN

# Effect of L-menthol on breathlessness and exercise capacity in COPD: a randomized crossover trial

Study code: Ment-COPD Date: 2025-11-17

NCT number: NCT05888597 Sponsor: Region Skåne, Represented by

Pia Malmqvist Lung- och allergikliniken, SUS Lund

Principal Investigator Zainab Ahmadi

Pulmonary physician

## **Statistical Analysis Plan**

The **primary outcome** is the post-dose difference in breathlessness intensity ratings during exercise at isotime, defined as the highest equivalent 1-minute interval of exercise completed by a given participant during each constant-load CPET. The **co-primary outcome** is the post-dose difference in exercise endurance time (EET), defined as the duration of loaded pedaling during constant-load CPET. Secondary outcomes include additional physiological and perceptual responses assessed at isotime and at peak exercise (end of test).

#### **Data Presentation:**

- Normally distributed continuous variables will be expressed as mean  $\pm$  standard deviation (SD).
- Skewed continuous variables will be expressed as median with range or interquartile range (IQR).
- Categorical variables will be presented as frequencies and percentages.

## **Comparisons:**

- Baseline characteristics will be compared using independent t-tests (continuous normal), Wilcoxon rank-sum tests (continuous non-normal), and chi-square tests (categorical).
- For CPET outcomes, within-subject comparisons between menthol and placebo will be performed using paired t-tests for normally distributed variables and Wilcoxon signed-rank tests for non-normal variables. Categorical outcomes will be analyzed using McNemar's test.
- CPET variables will be compared between conditions at isotime and peak exertion.

### Modeling:

Changes during CPET may be further analyzed using mixed-effects regression models to account for repeated measures.

#### Reporting:

Estimates will be presented as mean differences (menthol minus placebo) with 95% confidence intervals (CIs). Statistical significance will be defined as two-sided p < 0.05.

#### **Software:**

Analyses will be conducted using Stata (StataCorp LP; College Station, TX) [or specify alternative if applicable].

## **Figures**

Figures will be adapted from Abdallah et al. (2017) to illustrate perceptual and physiological responses during constant-load exercise testing. These will include:

- Panels a–c: Symptom ratings (breathlessness intensity, breathlessness unpleasantness, and leg discomfort) plotted against time during exercise for menthol and placebo conditions.
- Panels d-f: Post-dose differences (menthol minus placebo) at isotime and peak exercise for breathlessness intensity, unpleasantness, and exercise endurance time (EET), including individual participant data and group means with 95% CIs.
- **Panels g–i:** Distribution of individual responses and indication of clinically meaningful thresholds (e.g., minimally clinically important difference).

These figures will visualize symptom trajectories, treatment effects, and variability across participants, highlighting both statistical and clinical significance.

Figure 1: CONSORT diagram showing the flow of participants through each stage of the study



Table 1: Baseline participant characteristics (t-test for continuous variables with normal distribution, ranksum test for continuous non-normal variables and chi-

square for categorical variables).

| square for categorical variables). | | | 1 |
|---|---|---|---|
| Parameter | Menthol first | Placebo first | All participants |
| N (%) | | | |
| Male:female (n) | | | |
| Age, mean years (SD) | | | |
| Height (cm) | | | |
| Weight (kg) | | | |
| BMI kg/m <sup>2</sup> , mean (SD) | | | |
| Smoking history, pack-years (SD) | | | |
| Physical activity during normal week | | | |
| Thy stour west they warming mornion week | | | |
| Post-bronchodialator pulmonary | | | |
| function (spirometry) | | | |
| FEV1, L (SD) | | | |
| FEV <sub>1</sub> ,% predicted (SD) | | | |
| FVC, L (SD) | | | |
| FVC, % predicted (SD) | | | |
| FEV <sub>1</sub> /FVC, L (SD) | | | |
| FEV <sub>1</sub> /FVC, % of predicted (SD) | | | |
| Breahlessness and health status | | | |
| mMRC 0-4 | | | |
| CAT total Score | | | |
| CAT breathlessness | | | |
| CAT activity limitation | | | |
| MDP A1 total | | | |
| Dyspnea 12 | | | |
| Dyspnea severity likert | | | |
| SF12 q1 – q12 | | | |
| Change between visit 1 and 2 (GIC- | | | |
| scale) | | | |
| Change between visit 2 and 3 (GIC- | | | |
| scale) | | | |
| TI I I I | | | |
| Underlying conditions | | | |
| Ischaemic heart disease | | | |
| Angina Pectoris | | | |
| AF | | | |
| Heart failure | | | |
| Hypertension | | | |
| Hyperlipidemia | | | |
| Diabetes | | | |

| Obstructive sleep apnea | | |
|----------------------------------------|---|---|
| Asthma | | |
| Other lung disease | | |
| Tuberculosis | | |
| Rheumatic disease | | |
| Stroke | | |
| Cancer | | |
| Depression or anxiety | | |
| None | | |
| Other | | |
| Other | | |
| Medications | | |
| Diuretics | | |
| Beta blocker | | |
| Calcium antagonist | | |
| Renin-angiotensin system blocker | | |
| Insulin | | |
| Other diabetic medication | | |
| Anti hyperlipidemic drug | | |
| Inhalators for COPD/asthma | | |
| Anticoagulants | | |
| Antidepressants/anxiolytics | | |
| Sleep medication or other | | |
| benzodiazepines | | |
| Other | | |
| COPD medication | | |
| LABA+LAMA | | |
| LABA+LAMA+ICS | | |
| LABA | | |
| LAMA | | |
| LABA+LAMA+Daxas | | |
| LABA+LAMA+ICS+Daxas | | |
| Physiological responses at incremental | | |
| cycle test (visit 1) | | |
| Cycle exercise time (min) | | |
| Workload, W | | |
| Workload, % of predicted | | |
| Heart rate, beats/min | | |
| Breathing frequency (breaths/min) | | |
| SpO <sub>2</sub> (%) | | |
| V <sub>O2</sub> , mL/kg/min, | | |
| $V_{O2}$ (% of predicted), | | |
| V'CO2 (ml/kg/min) | | |
| , coz (mingimm) | l | L |

| RER |
|-----------------------------------------|
| V' <sub>E,</sub> L/min |
| $V_{T}$ , L |
| V'E/V'CO2 |
| Perceptual responses during test (visit |
| 1) |
| Breathlessness intensity, Borg units |
| Breathlessness discomfort, Borg units |
| Leg discomfort, Borg units |
| Reasons for stopping exercise (visit 1) |
| Breathlessness (n) |
| Leg discomfort (n) |
| Breathlessness and Leg discomfort (n) |
| Breathlessness ratings after test |
| (visit 1) |
| MDP (A1 + dimensions) |
| D12 |
| Self-reported motivation for |
| completing test (visit 1) |

**Table 2:** Effect of menthol versus placebo on physiological and perceptual responses at a standardized submaximal time during constant-load exercise testing (isotime) and at the symptom limited peak of constant-load exercise testing among individuals with Chronic obstructive pulmonary disease. (t-test for continuous variables with normal distribution, ranksum test for continuous non-normal variables and chi-square for categorical

variables). (Visit 2 and 3)

| Parameter, | t 2 and 3) Rest | | | Isotime | | | Peak | | |
|---|---|---|---|---|---|---|---|---|---|
| mean (SD) | 126 (1.11 12) | | | | | | | | |
| | Menthol | Placebo | Mean<br>difference<br>(95% CI) | Menthol | Placebo | Mean<br>difference<br>(95% CI) | Menthol | Placebo | Mean<br>difference<br>(95% CI) |
| Physiological | | | | | | , | | | , |
| responses | | | | | | | | | |
| Cycle exercise | | | | | | | | | |
| time, min | | | | | | | | | |
| Heart rate, | | | | | | | | | |
| beats/min | | | | | | | | | |
| Breathing | | | | | | | | | |
| frequency, | | | | | | | | | |
| breaths/min | | | | | | | | | |
| SpO2, % | | | | | | | | | |
| V' <sub>O2,</sub> ml/kg/min | | | | | | | | | |
| V' <sub>O2,</sub> % of | | | | | | | | | |
| predicted | | | | | | | | | |
| V' <sub>CO2</sub> | | | | | | | | | |
| (ml/kg/min) | | | | | | | | | |
| RER | | | | | | | | | |
| V' <sub>E</sub> , L/min | | | | | | | | | |
| $V_{T,L}$ | | | | | | | | | |
| V'E/V'CO2 | | | | | | | | | |
| PETH CO2 | | | | | | | | | |
| Perceptual | | | | | | | | | |
| responses | | | | | | | | | |
| Breathlessness | | | | | | | | | |
| intensity (Borg | | | | | | | | | |
| CR10) | | | | | | | | | |
| Breathlessness | | | | | | | | | |
| unpleasantness | | | | | | | | | |
| (Borg CR10) | | | | | | | | | |
| Leg discomfort | | | | | | | | | |
| (Borg CR10) | | | | | | | | | |
| Significant | | | | | | | | | |
| breathlessness | | | | | | | | | |
| (>2, n (%) | | | | | | | | | |
| Reasons for | | | | | | | | | |
| stopping test | | | | | | | | | |
| Breathlessness | | | | | | | | | |
| (n) | | | | | | | | | |
| Leg discomfort | | | | | | | | | |
| (n) | | | | | | | | | |

| Breathlessness |
|----------------|
| and Leg |
| discomfort (n) |
| Level of self- |
| reported |
| motivation |
| Breathlessness |
| ratings after |
| tests |
| MDP |
| Dyspnea 12 |

Mean differences are for menthol minus placebo.

## Figures:



FIGURE 2 Effect of immediate-release oral morphine *versus* placebo on exertional breathlessness and exercise endurance in adults with advanced chronic obstructive pulmonary disease (COPD) and chronic breathlessness syndrome. Mean±sem a) breathlessness intensity ratings, b) breathlessness unpleasantness ratings and c) leg discomfort ratings at rest and during constant-load cycle exercise testing at 75% of peak incremental power output. Individual participant post-dose values and post-dose differences in d and g) breathlessness intensity ratings during exercise at isotime, e and h) breathlessness unpleasantness ratings during exercise at isotime and f and i) exercise endurance time, where red symbols with dashed horizontal lines in panels d, e and f) denote mean±sem. Dashed horizontal lines in panels g and i denote minimally clinically important difference for breathlessness intensity [36] and exercise endurance time [37].  $\Delta$ : post-dose difference (*i.e.*, morphine *minus* placebo). \*: p<0.05 *versus* placebo.

Example from Abdallah 2017 - panels (a,b och c) to be reported for each of "intensity,unpleasantness and leg discomfort". To be presented as the above example but change "Morphine" to "Menthol".